CLINICAL TRIAL: NCT02510534
Title: A Prospective Randomized Trial to Study the Effect of Luteal Progesterone Support on Pregnancy Rates in Combined Clomiphene Citrate and Gonadotropin Ovulation Induction Protocol With Intrauterine Insemination.
Brief Title: Effect of Luteal Progesterone Support on Pregnancy Rates With Combined Clomid/ Gonadotropin & IUI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: unable to enroll participants who meet the criteria
Sponsor: Northwest Center for Infertility and Reproductive Endocrinology (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVFFL001v2
Record Dates: First submitted 2015-07-24; First posted 2015-07-29 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Pregnancy
MeSH Terms: interventions — Gonadotropins; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): This arm receives Menopur 150 international units x 1 dose
  Interventions: Drug: Menopur 150 international units
- Treatment (Active Comparator): This arm receives Menopur 150 international units x 1 dose and Endometrin 100mg twice a day x 14 days
  Interventions: Drug: Menopur 150 international units; Drug: Endometrin 100 mg

INTERVENTIONS:
Drug: Menopur 150 international units — Menopur 150 international units given x 1 dose
  Other Names: Gonadotropin
Drug: Endometrin 100 mg — Endometrin 100mg twice daily x 14 days
  Other Names: Progesterone
  Arms: Treatment

SUMMARY:
To determine the difference in clinical pregnancy rates with and without luteal progesterone support in a young reproductive aged population having undergone ovulation induction with combined clomiphene citrate and gonadotropin protocol with intrauterine insemination.

DETAILED DESCRIPTION:
To determine the difference in clinical pregnancy rates with and without luteal progesterone support in a young reproductive aged population having undergone ovulation induction with combined clomiphene citrate and gonadotropin protocol with intrauterine insemination.

Patients will be randomized in a treatment arm or control arm. The treatment arm receives the luteal progesterone support and the control arm does not. Each arm will have 260 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-37
* BMI 19-34 kg/m2
* Day 2-3 Follicle stimulating hormone (FSH) less than 10IU/mL
* Estradiol (E2) less than 80 pg/mL
* Anti-mullerian hormone (AMH) more than 1.5 ng/mL; or antral follicle count (AFC) up to 10
* Two patent fallopian tubes confirmed by hysterosalpingogram (HSG) or chromopertubation
* Normal uterine cavity confirmed by HSG, saline sonohysterogram (SIS) or hysteroscopy

Exclusion Criteria:

* Severe male factor (total count less than 10 million sperm)
* Systemic diseases not limited to diabetes
* Pregnancy within 3 months
* More than 1 prior cycle of gonadotropin treatment
* Any ovarian cyst >15mm that has persisted for > 1 month
* Endometrioma and/or Endometriosis-stage III or IV
* Submucosal uterine fibroids; untreated endometrial polyps >1 cm;abnormal reproductive tract bleeding
* Intolerance or allergy to study drug
* Substance abuse (including alcohol and tobacco)
* History of chemotherapy (except for gestational conditions) or radiotherapy
* Minors and those adults not capable of consenting on their own

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 520 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Effect on Pregnancy rate measured by detectable embryonic cardiac activity | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Christie, MD, Principal Investigator — IVF FL
Locations (1):
- Ivf Florida, Margate, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided